CLINICAL TRIAL: NCT02966626
Title: Dapaglifozin in Type 2 Diabetes Mellitus Patients: A Single-centre Retrospective Cohort Study
Brief Title: A Real World Experience of Dapagliflozin in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: 20163-2261
Record Dates: First submitted 2016-11-14; First posted 2016-11-17 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Type2 Diabetes
Keywords: Pragmatic, Sodium-Glucose Transporter 2 inhibitor, Malaysia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Type 2 diabetes mellitus (T2DM) is creating a health pandemic globally. Management of type 2 diabetes involves combination of lifestyle intervention and drug intervention, which includes sodium-glucose transporter 2 (SGLT-2) inhibitors, such as dapagliflozin. Dapagliflozin (Forxiga®) was approved by the Malaysian Drug Authority for the treatment of type 2 diabetes in 2014. This study will describe the characteristics of patients who are prescribed dapagliflozin by diabetologists/endocrinologists in a tertiary referral center and describe their glycaemic control, weight, and renal function at baseline and during use of dapagliflozin.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes among adults >18 years old is 17.5% in Malaysia, where half of them are undiagnosed. Diabetes also accounts for 14.5% of all-cause mortality worldwide, with close to half of the deaths are in subjects <60 years old. These highlight the importance of early diagnosis of disease, timely intervention with appropriate therapy, and treating type 2 diabetes patients to goal to prevent the development of complications.

Asian type 2 diabetes phenotypes are different than Caucasians, i.e. significant pancreatic beta-cell dysfunction, higher visceral adiposity, more vulnerable to cardio-renal complications. Although clinical trials of SGLT-2 inhibitors have been published, real-world data on the use of this new class of antidiabetic medication is still lacking, in particularly among Asians.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM prior to the first prescription of dapagliflozin
* Patients with T2DM who are initiated with dapagliflozin from March 2014 till December 2015
* Patients need to be on dapagliflozin therapy for at least six consecutive months from the index date
* Patients need to have diabetologists/endocrinologists' follow up for at least six months after the initiation of dapagliflozin

Exclusion Criteria:

* Patients with T2DM who are initiated with dapagliflozin after December 2015
* Patients with incomplete electronic medical records
* Patients with Type 1 diabetes
* Patients with latent autoimmune diabetes of adults (LADA)
* Female Patients with T2DM who are found to be pregnant during the treatment period of dapagliflozin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult T2DM patients who received at least one prescription for dapagliflozin for the first time between March 2014 and December 2015 at the University of Malaya Medical Center (UMMC) will be recruited. UMMC is an academic medical institution with 1,300 beds, serving a population of 1.8 million in Kuala Lumpur, Malaysia.
  The date of the first prescription for dapagliflozin in the Hospital Pharmacy Database is defined as the index date. Dapaglifozin is only available at the study site from March 2014 onwards.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months
  To assess the change in HbA1c from baseline to 6 months

SECONDARY OUTCOMES:
Change in body weight | 6 months
  To assess the change in body weight from baseline to 6 months
Change in estimated glomerular filtration rate | 6 months
  To assess the change in estimates glomerular filtration rate from baseline to 6 months
Change in albuminuria | 6 months
  To assess the change in albuminuria from baseline to 6 months
Change in body mass index | 6 months
  To assess the change in body mass index from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ling LIM, MRCP (UK), Principal Investigator — University of Malaya, Malaysia

IPD SHARING:
Plan to Share IPD: No